CLINICAL TRIAL: NCT02861976
Title: Screening in Trauma for Opioid Misuse Prevention (STOMP): Screen Development and Pilot Implementation Study
Brief Title: Screening in Trauma for Opioid Misuse Prevention
Acronym: STOMP
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-0430; 3152 (Other: Study Team); A532050 (Other: UW Madison); SMPH/FAMILY MEDICINE/CL-WINGRA (Other: UW Madison); Protocol Version 9/5/2019 (Other: UW Madison)
Record Dates: First submitted 2016-02-09; First posted 2016-08-10 (Estimated); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Opioid risk screen development & implementation — Development of a screening tool for the risk of opioid misuse in patients with traumatic injury.

SUMMARY:
The current study seeks to begin the crucial work of creating effective protocols to prevent opioid misuse, addiction, and related complications by developing and pilot testing an opioid risk screening protocol at Wisconsin trauma centers.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient victim of traumatic injury
* Expected need for post-discharge outpatient opioid analgesia
* English speaking
* Disposition to short-term rehabilitation facility is allowed

Exclusion Criteria:

* Disposition to a skilled nursing or long-term acute care facility
* Current active opioid use disorder or current active participation in a program of recovery for another substance use disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of UW Trauma Inpatient Service with expected need for post discharge with outpatient opioid analgesia.
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Opioid use disorder (CIDI-SAM) or opioid misuse (COMM) Opioid Use Disorder in 6 Months Post Traumatic Injury | 6 months subject participation
  This data will be analyzed in tandem with patient demographics, physical and mental health, and hypothesized risk factors for opioid misuse.

CONTACTS AND LOCATIONS:
Overall Officials: Randall Brown, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brown R, Deyo B, Riley C, Quanbeck A, Glass JE, Turpin R, Hetzel S, Nicholas C, Cruz M, Agarwal S. Screening in Trauma for Opioid Misuse Prevention (STOMP): study protocol for the development of an opioid risk screening tool for victims of injury. Addict Sci Clin Pract. 2017 Dec 4;12(1):28. doi: 10.1186/s13722-017-0097-6. PMID 29198186